CLINICAL TRIAL: NCT05466981
Title: Smoking Cessation Intervention for Persons Infected With Hepatitis C Virus
Brief Title: HCV-Smoking Cessation Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Prisma Health-Upstate (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 00103095
Record Dates: First submitted 2021-07-26; First posted 2022-07-20 (Actual); Last update posted 2022-07-20 (Actual); Status verified 2021-07

CONDITIONS: Hepatitis C; Smoking Cessation
MeSH Terms: conditions — Hepatitis C; Smoking Cessation

STUDY DESIGN:
Intervention Model Description: We conducted a single-arm pilot study in order to test the feasibility and preliminary efficacy of a smoking cessation intervention for people with HCV while they received standard of care treatment: antiviral medication and provider/laboratory visits.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Current smokers with an HCV infection (Experimental): Persons who currently smoke cigarettes and are also HCV RNA+
  Interventions: Behavioral: Cognitive Behavioral Counseling

INTERVENTIONS:
Behavioral: Cognitive Behavioral Counseling — The intervention consisted of 12 weeks of HCV treatment combined with smoking cessation pharmacotherapy and brief behavioral counseling conducted by a LMSW. The brief behavioral counseling consisted of cognitive behaioral components and was provided by phone and in-person. The intervention followed these 5 phases: increase motivation to quit smoking, quit attempt, maintain short-term abstinence, and lapse and relapse prevention.

SUMMARY:
A 12-week study for patients who are being treated for Hepatitis C and would like to quit smoking. During the 12 weeks of Hepatitis C treatment, the research team will have counseling sessions with the participants to discuss challenges related to Hepatitis C and smoking.

DETAILED DESCRIPTION:
A 12-week smoking cessation intervention addressing concurrently HCV and smoking cessation The Standard of care for HCV is 12 weeks of oral medication with 3 in-person provider/laboratory visits throughout. This study utilizes both in-person and phone counseling and health education sessions. Each session will address a different topic related to HCV, smoking, and how both smoking and HCV affect health and quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Adults (≥18 years old)
* Current HCV infection (HCV RNA+)
* Current cigarette smoking
* Patients in contemplation / preparation stage of change

Exclusion Criteria:

* Inability to speak/read English, as materials will be provided in English
* Current suicidal ideation as determined by the PHQ-9, requiring a greater level of clinical care
* Severe medical or psychiatric disability that prevents participant from ability to comprehend or consent to study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2020-11-23 (Actual); Primary Completion 2021-11-11 (Actual); Study Completion 2021-11-11 (Actual)

PRIMARY OUTCOMES:
Change in the number of cigarettes smoked per day (CPD) | baseline (week 0) to end of treatment (week 12)
  We will track the number of cigarettes the participant smokes per day at each weekly visit, then compare the CPD at baseline during week 0 to the end of treatment at week 12.
Change in Fagerstrom Test for Nicotine Dependence (FTND) score | baseline (week 0) to end of treatment (week 12)
  We will calculate the participant's FTND score at the baseline visit during week 0 and compare it to their FTND score at the end of treatment visit during week 12.

SECONDARY OUTCOMES:
Change in depressive symptomology using Patient Health Questionnaire (PHQ-9) score | baseline (week 0) to end of treatment (week 12)
  We will calculate the participant's PHQ-9 score at the baseline visit during week 0 and compare it to their PHQ-9 score at the end of treatment visit during week 12.
Number of quit attempts | baseline (week 0) to end of treatment (week 12)
  We will measure the number of quit attempts made throughout the intervention from baseline to end of treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Irene Pericot-Valverde, PhD, Principal Investigator — Prisma Health; Alain Litwin, MD, Study Director — Prisma Health
Locations (1):
- Prisma Health Internal Medicine Clinic, Greenville, South Carolina, United States

IPD SHARING:
Plan to Share IPD: No